CLINICAL TRIAL: NCT05915403
Title: The Effect of Frequency of Sexual Intercourse on Symptoms in Women With Fibromyalgia
Brief Title: Frequency of Sexual Intercourse,Women With Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savaş Karpuz, Medical doctor, Konya Beyhekim Training and Research Hospital
Other Study IDs: 2021-01-05
Record Dates: First submitted 2023-06-12; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Fibromyalgia; Pain; Depression
MeSH Terms: conditions — Fibromyalgia; Pain; Depression | interventions — Visual Analog Scale

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: female patient with fibromyalgia
  Interventions: Diagnostic Test: Fibromyalgia Impact Questionnaire
- healthy controls: women

INTERVENTIONS:
Diagnostic Test: Fibromyalgia Impact Questionnaire — diagnostic tests
  Other Names: Visual Analog Scale; Beck Depression Inventory; Widespread Pain Index; Symptom Severity Scale; frequency of sexual intercourse
  Groups: Patient

SUMMARY:
Does frequency of sexual intercourse affect symptom severity in female patients with fibromyalgia?

ELIGIBILITY:
Inclusion Criteria:

* Female patient with fibromyalgia

Exclusion Criteria:

* Uncontrollable systemic disease (cardiovascular, pulmonary, hepatic, renal, hematological),
* Major psychiatric disease,
* Endocrine disease,
* Pregnancy
* Menopausal status,
* Antihypertensive, antidepressant, anxiolytic, antiepileptic drugs use

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: tertiary healthcare facility
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 1 week
  pain level 0-10, higher scores indicate worse outcome
frequency of sexual intercourse | 3 mounths
  mean monthly frequency of sexual intercourse in the last 3 months
Fibromyalgia Impact Questionnaire | 1 week
  0-80, higher scores indicate worse outcome

SECONDARY OUTCOMES:
Beck Depression Inventory | 1 week
  0-63, higher scores indicate worse outcome
Widespread Pain Index | 1 week
  0-19, higher scores indicate worse outcome
Symptom Severity Scale | 1 week
  0-12, higher scores indicate worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Beyhekim Research and Training Hospital, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Maunder L, Schoemaker D, Pruessner JC. Frequency of Penile-Vaginal Intercourse is Associated with Verbal Recognition Performance in Adult Women. Arch Sex Behav. 2017 Feb;46(2):441-453. doi: 10.1007/s10508-016-0890-4. Epub 2016 Nov 14. PMID 27844312
- [Result] Blaicher W, Gruber D, Bieglmayer C, Blaicher AM, Knogler W, Huber JC. The role of oxytocin in relation to female sexual arousal. Gynecol Obstet Invest. 1999;47(2):125-6. doi: 10.1159/000010075. PMID 9949283
- [Result] Burleson MH, Trevathan WR, Todd M. In the mood for love or vice versa? Exploring the relations among sexual activity, physical affection, affect, and stress in the daily lives of mid-aged women. Arch Sex Behav. 2007 Jun;36(3):357-68. doi: 10.1007/s10508-006-9071-1. PMID 17109236
- [Result] Ainsworth BE, Haskell WL, Herrmann SD, Meckes N, Bassett DR Jr, Tudor-Locke C, Greer JL, Vezina J, Whitt-Glover MC, Leon AS. 2011 Compendium of Physical Activities: a second update of codes and MET values. Med Sci Sports Exerc. 2011 Aug;43(8):1575-81. doi: 10.1249/MSS.0b013e31821ece12. PMID 21681120